CLINICAL TRIAL: NCT03814083
Title: Effects of Transcranial Direct Current Stimulation for Enhancing Cognitive Function in Children With Autism Spectrum Disorder
Brief Title: Transcranial Direct Current Stimulation in Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Yvonne Han, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20171230001
Record Dates: First submitted 2019-01-11; First posted 2019-01-23 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Transcranial Direct Current Stimulation; Autistic Disorders Spectrum; Electroencephalography
MeSH Terms: conditions — Child Development Disorders, Pervasive | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active-tDCS and Sham-tDCS (Experimental): For active-tDCS condition, participants will receive stimulation on the dorsolateral prefrontal cortex with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds. Following that, a twenty-minute executive functional training task will be initiated five minutes subsequent to the stimulation mode, and the stimulation will be terminated when the training task ends. On the other hand, for sham-tDCS condition, participants will receive initial stimulation with ramp up and ramp down mode for 30 seconds, eliciting a tingling sensation on the scalp then it will be discontinued. Participant will also receive the twenty-minute executive functional training task five minutes subsequent to the stimulation mode.
  Interventions: Device: Active-tDCS; Device: Sham-tDCS
- Active-tDCS and wait-list (Active Comparator): For active-tDCS condition, participants will receive stimulation on the dorsolateral prefrontal cortex with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds. Following that, a twenty-minute executive functional training task will be initiated five minutes subsequent to the stimulation mode, and the stimulation will be terminated when the training task ends. On the other hand, participants in the wait-list control group will not receive any intervention.
  Interventions: Device: Active-tDCS; Other: Wait-list
- Sham-tDCS and wait-list (Sham Comparator): For sham-tDCS condition, participants will receive initial stimulation with ramp up and ramp down mode for 30 seconds, eliciting a tingling sensation on the scalp then it will be discontinued. Participant will also receive the twenty-minute executive functional training task five minutes subsequent to the stimulation mode. On the other hand, participants in the wait-list control group will not receive any intervention.
  Interventions: Device: Sham-tDCS; Other: Wait-list

INTERVENTIONS:
Device: Active-tDCS — Active-tDCS over 10 sessions in 2 weeks (once per day, for 10 consecutive working days), while performing the executive function training tasks. Also, participants will complete an online cognitive training program while they receive active tDCS stimulation for 10 training sessions. The training session will last for 20 minutes and the online cognitive training program is comprised of 5 exercises targeting at information processing speed and executive function capacities. Each exercise lasts for approximately 4 minutes, totaling approximately 20 minutes.
  Arms: Active-tDCS and Sham-tDCS; Active-tDCS and wait-list
Device: Sham-tDCS — Sham-tDCS stimulation over 10 sessions in 2 weeks (once per day, for 10 consecutive working days), while performing the executive function training tasks. Also, participants will complete an online cognitive training program while they receive sham-tDCS stimulation for 10 training sessions. The training session will last for 20 minutes and the online cognitive training program is comprised of 5 exercises targeting at information processing speed and executive function capacities. Each exercise lasts for approximately 4 minutes, totaling approximately 20 minutes.
  Arms: Active-tDCS and Sham-tDCS; Sham-tDCS and wait-list
Other: Wait-list — No intervention
  Arms: Active-tDCS and wait-list; Sham-tDCS and wait-list

SUMMARY:
Background: Transcranial Direct Current Stimulation (tDCS) is a form of non-invasive brain stimulation that has aroused increased interests in the past decade. Not only that it is transient with little side-effects, and can be well-tolerated by children, it is also affordable and readily accessible, making it an appealing treatment option for autism spectrum disorder (ASD).

Objective: (1) To assess the therapeutic effects of tDCS when combined with cognitive training for 10 consecutive weekdays on improving cognitive processing in adolescents with ASD, relative to control group receiving sham-stimulation, and (2) to evaluate the associated neural mechanisms underlying the treatment effect of tDCS on adolescents with ASD.

Methods: 105 adolescents with ASD will be randomly assigned to active- (n=35), sham- (n=35) tDCS, or no-treatment control (n=35) groups. Twenty minute sessions of 1 mA cathodal stimulation to the left dorsolateral prefrontal cortex (DLPRC) in conjunction with cognitive training exercise will be provided on 10 consecutive weekdays. EEGs, functional near-infrared spectroscopy, and neuropsychological tests will be administered before, 1 day and 6 months after the series of tDCS sessions.

Hypothesis: We hypothesized that cathodal (inhibitory) tDCS over the left DLPRC will induce (1) stimulation-linked facilitation of learning and enhanced processing speed and resultant improvement of cognitive functioning, in executive function, relative to the sham-tDCS and the wait-list controls, (2) active-tDCS, but not sham-tDCS and wait-list controls, will modulate the intra- and inter-hemispheric neural connectivity, indexed by altered level EEG theta coherence and aberrant fNIRS haemodynamic measures, across brain areas implicated in executive functioning.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a lifelong neurodevelopmental disorder characterized by disturbances in communication, poor social skills, and aberrant behavior. ASD often causes considerable emotional and financial stress on the patients, their families and the community. Prevalence of ASD is high, with recent statistics reported at one in 68. Thus far, there is no cure for ASD and the disorder remains a highly disabling condition in spite of the existing treatment options. Hence, more effective novel therapeutic approaches are urgently needed. In the past 10 years, transcranial direct current stimulation (tDCS), a brain stimulation technique, has been intensively investigated regarding its physiologic mechanisms of action render empirical support of its application in clinical setting.

Cognitive and social deficits in ASD. Individuals with ASD often appear rigid and inflexible, show a strong liking for repetitive behaviour and elaborate rituals. One reason for the aberrant behaviour in ASD may be attributed to their deficient processing speed and resultant cognitive deficits. Slow processing speed relates to a reduced capacity of executive function to recall and formulate thoughts and actions automatically, with the result that autistic individuals with slow processing speed would have great difficulty learning or perceiving the relationships across multiple experiences. As a result, these individuals compensate for the impaired ability to integrate information from the environment by memorizing visual details or individual rules from each situation. This explains why individuals with the disorder tend to follow routines in precise details and show great distress with trivial changes in the environment.

Disordered functional connectivity underlies cognitive dysfunction in ASD: Neural connectivity problem has been widely reported in individuals with ASD. For example, diffusion tensor imaging (DTI) and Electrophysiological studies have reported reduced myelin integrity in the ventromedial prefrontal cortex and at the temporoparietal junctions. Similarly, functional imaging studies have found reduced synchronization between activated brain areas on tests of working memory, executive function, and interpretations of the affective meaning of actions in individuals with ASD.

Cortical inhibition and excitability (E/I ratio) in ASD: The significantly variability in symptom presentation in ASD can now be understood as a manifestation of a neural systems disorder, with abnormalities found in the interaction among different brain areas attributable to some brain connectivity disorder. Related to the underlying connectivity problem in ASD is the dysregulation of cortical excitability. One emerging principle is that the cognitive deficits in autism are caused by excessively high level of excitation within the neural circuits that mediate the different cognitive functions in ASD. The suggested role of the increased ratio of cortical cellular excitation to inhibition (E/I balance) in the pathophysiology of of ASD is supported by recent studies which have shown that a reduction in GABAergic signalling is a common feature in the brains of autistic individuals, with enhancement of excitatory glutamatergic signalling as the underlying mechanism. These findings are consistent with neural connectivity studies suggesting that cortical cellular E/I imbalance or hyper-excitability could disrupt the normal progressive differentiation and elaboration of functional connectivity in the developing brain.

Effects of Transcranial Direct Current Stimulation (tDCS) on modulating cortical excitation/inhibition balance: tDCS is a non-invasive neuromodulation method which influences cortical activity level, by applying low direct currents to the scalp through anodal and cathodal electrodes. Magnetic resonance spectroscopy (MRS) studies have reported that anodal tDCS increases cortical excitability by reducing local concentrations of the inhibitory neurotransmitter gamma-aminobutyric acid (GABA), whereas cathodal tDCS decreases cortical excitability by reducing excitatory glutamate levels. As cathodal tDCS can reduce cortical excitability caused by neuronal hyperpolarization, it is reasonable to assume that cathodal stimulation can be beneficial in ASD by decreasing the cortical excitability in the affected individuals with the disorder.

Therapeutic effect of tDCS on improving cognitive function: In the past decade, there has been a growing interest in studying the effect of tDCS to alter various central nervous system functions, including motor control, attention, memory, language, and emotion, and to modulate brain activity level and functional connectivity in healthy and patient population. To date, more than 100 tDCS studies have shown promising results and reported instant tDCS-induced positive effects on cognitive functions, without any safety problem or adverse side-effect. Additionally, synaptically driven aftereffects were induced with sufficient tDCS duration. It has been shown that a single-session of tDCS for 10-13 minutes could induce an hour of after-effect, and 10 repeated sessions of tDCS coupled with therapeutic task in children with perinatal stroke were associated with changes in spectroscopic biomarkers 1 week after stimulation and sustained clinical improvement at a 2-month follow-up visit. Interestingly, more significant behavioral/cognitive improvement have been reported when tDCS were paired with therapeutic task than receiving tDCS alone. These findings are consistent with the notion that performing therapeutic task during tDCS can direct the stimulation effect to the neural circuits involved. In which, the coupling of tDCS with therapeutic task can enhance learning through inducing long term potentiation-changes to underlying brain regions and modulates brain activity associated with the task. This in turn can lead to greater synaptic modification and improved task performance. Among the various tDCS protocols, stimulation on the dorsolateral prefrontal cortex (DLPFC) is one of the widely applied montages. tDCS over the DLPFC has been shown to improve cognitive functions such as working memory, inhibitory control, emotional state and processing in neuropsychiatric patients.

Although these preliminary findings in neuropsychiatric patients are encouraging, empirical studies on the application of tDCS on individuals with ASD are limited. The research that has been performed, however, is encouraging. For example, one clinical case study of autistic patient who received 10 consecutive daily 20-min sessions of 1.5mA cathodal tDCS over the left DLPFC, showed persisted significant improvement in his highly disabling behavioural symptoms at a 3-month follow-up visit. Additionally, tDCS over the left DLPFC has also been shown to modulate inhibitory control of behavioural outbursts and language acquisition in minimally verbal children with ASD. Given the promising outcomes of brain stimulation treatment of resistant neuropsychiatric disorders, the present study thus aims to explore the repetitive effect of tDCS on improving cognitive functions, with particular interest in enhancing functional connectivity, in adolescents with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are confirmed by a clinical psychologist based on the Diagnostic and Statistical Manual of Mental Disorders-5th Ed (DSM-V) criteria of Autism spectrum disorder and structured interview with their parents or primary caregivers on their developmental history using the Autism Diagnostic Interview-Revised (ADI-R).
* Individuals with intelligence quotient above 70
* Individuals who demonstrate the ability to comprehend testing and stimulation instructions

Exclusion Criteria:

* Individuals with severe motor dysfunctions that would hinder their participation, and those with history of other neurological and psychiatric disorders and head trauma, or on psychiatric medication will be excluded from the study

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in behavioral measures - Early Adolescent Temperament Questionnaire - Revised - Effortful control subscale (EATQ-R-EC) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  EATQ-R-EC is an 18-item self-rated questionnaire composed of 3 sub-components under effortful control, namely attentional control, inhibitory control and activation control.
Change in behavioral measures - Autism Quotient (AQ) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  AQ serves as a screening test for autism spectrum disorders. Given its sensitivity to subtle autistic features, it is thus adopted in present study to rule out possibilities of children having unidentified autism. The questionnaire is rated on a 4-point Likert scale, from 0 (definitely agree) to 3 (definitely disagree) on a total of 50 items. Higher scores suggest greater severity level of autistic features.
Change in behavioral measures - Social Responsiveness Scales (SRS) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  SRS-2 for measures participants' social communication abilities that are highly related to frontal lobe dysfunction. It is a 4-point scale tapping on the aspects of social awareness, social cognition, social communication, social motivation, and restricted interests and repetitive behavior. Higher scores indicate greater difficulties in socialization.
Change in CANTAB® cognitive test - Stop Signal Task (SST) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  Cambridge Neuropsychological Test Automated Battery (CANTAB®) includes computerized tests correlated to neural networks and have demonstrated high sensitivity in detecting changes in neuropsychological performance. SST assesses a participants' motor inhibition of a prepotent response. The participant is required to respond to an arrow stimulus by selecting one of two options, depending on the direction in which the arrow points. If an audio tone is present, the subject must withhold making the response.
Change in CANTAB® cognitive test - Reaction Time (RTI) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  RTI assesses motor and mental response speeds, reaction time, response accuracy and impulsivity. Participants are required to react as soon as a yellow dot appears on screen. Specifically, movement and reaction time will be measured, where shorter duration reflects faster processing speed.
Change in CANTAB® cognitive test - One Touch Stockings of Cambridge (OTS) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  OTS assesses the spatial planning ability. The participant is required to determine the number of steps required to move the balls such that the pattern copies the desired patterns (correct answer). The OTS comprises of 4 problem sets to reflect increasing demands on planning.
Change in CANTAB® cognitive test - Multitasking Test (MTT) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  MTT assesses the ability to resolve the interference of task-irrelevant information (stroop-like effect). The test displays an arrow which can appear on either the left or right side of the screen and can point to either the left or right side. In each trial, participants are presented with a cue that indicates which button to press according to two different rules. And the rules that participants have to follow may change from trial to trial in a randomized order. Participant's response latencies and error scores will be measured.
Change in CANTAB® cognitive test - Emotion Recognition Task (ERT) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  ERT assesses emotional recognition ability of an individual. The participant is required to determine the emotion of the face displayed from 6 options (i.e. sadness, happiness, fear, anger, disgust or surprise) after viewing the facial features of real individuals for 200 milliseconds.
Change in n-back task | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  The N-back paradigm consists of 0-back (i.e., low working memory load), 1-back (i.e., medium working memory load), and 2-back (i.e., high working memory load) conditions. For the 0-back condition, participants have to press the left button of a mouse when the digit "0" (i.e., target) appeared whereas to press the right button for occurrence of other digits. For 1-back condition, participants are required to press the left button when the presented digit was identical to the one presented in the previous trial (i.e., target), otherwise, press the right button. For 2-back condition, participants are required to press the left button when the presented digit was identical to the one presented two trials before (i.e., target), otherwise, press the right button. The accuracy rate and reaction time of each block across different conditions will be measured to reflect the capacity of working memory and processing speed.
Change in the Attention Network Task (ANT) | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  The computerized ANT paradigm measures different levels of attention network, namely alerting, orienting and conflicting monitoring. To measure alerting and/or orienting, 3 warning conditions will be presented - no-cue (baseline), center-cue (alerting) and spatial-cue (alerting plus orienting). Stimuli consisted of a row of 5 objects, with the object in the center being an arrow pointing either to the left or right, and 4 remaining objects being diamond-shaped stimuli. To assess conflict monitoring, the central arrow will be "flanked by congruent or incongruent stimuli". The target is flanked on either side by two arrows in the same direction (congruent) or in the opposite direction (incongruent). The participants are required to identify the direction of the arrow presented in the middle by pressing the left and right button respectively. Reaction times will be calculated to reflect subjects' performance.
Change in Electroencephalography (EEG) coherence measure | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  EEG coherence measure is a useful indicator of cortical connectivity between functional areas in the brain. It reflects the levels of synchronization between two cortical areas at different sites of the scalp. High coherence indicates a high level of synchronization between the two brain areas, whereas low coherence indicates a low level of synchronization. It has been shown that different EEG frequency bands correlate with different cognitive and emotional processes. EEG signals collected from the 19 electrode positions (Fp1, Fp2, F3, F4, F7, F8, Fz, T3, T4, T5, T6, C3, C4, Cz, P3, P4, Pz, O1, and O2) will be used.
Change in functional near-infrared spectroscopy (fNIRS) recording | First day of intervention,1 day and 6 months after the last day of intervention (3 time points)
  NIRS is a non-invasive neuroimaging procedure used to measure hemodynamic changes, in terms of oxyhemoglobin (HbO), deoxyhemoglobin (HbR) and total haemoglobin (HbT), associated with neuronal activities of the cerebral cortex in response to attending a task within a given period of time. In addition, functional connectivity will be measured, in which the synchronized responses to cognitive stimuli between and within the left and right frontal cortex will be computed in terms of zero lagged correlation. During the NIRS session, participants will be tested on the Attention Network Task (ANT), and the n-back task while their hemodynamic data are collected using the NIRS system.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Han, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

REFERENCES:
- [Derived] Han YMY, Chan MMY, Shea CKS, Lai OL, Krishnamurthy K, Cheung MC, Chan AS. Neurophysiological and behavioral effects of multisession prefrontal tDCS and concurrent cognitive remediation training in patients with autism spectrum disorder (ASD): A double-blind, randomized controlled fNIRS study. Brain Stimul. 2022 Mar-Apr;15(2):414-425. doi: 10.1016/j.brs.2022.02.004. Epub 2022 Feb 15. PMID 35181532